CLINICAL TRIAL: NCT00135759
Title: Place of Low-Dose Naltrexone in Opiate Detoxification
Brief Title: Addition of Naltrexone to Methadone Taper
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Paolo Mannelli, M.D., Duke University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-15469-1; R21-15469-1; DPMC
Record Dates: First submitted 2005-08-23; First posted 2005-08-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders; Substance-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Placebo Comparator): Drug
  Interventions: Drug: Placebo comparator
- 2 (Experimental): experimental
  Interventions: Drug: Naltrexone
- 3 (Experimental): experimental
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — low dose naltrexone in addition to daily methadone taper
  Arms: 2; 3
Drug: Placebo comparator — 1 capsule/day for 6 days
  Arms: Group 1
Drug: naltrexone — 0.125 mg capsule/day for 6 days
  Arms: 2
Drug: naltrexone — 0.250 mg capsule/day for 6 days
  Arms: 3

SUMMARY:
There is a continuing search for more effective opiate detoxification treatments. This study's purpose is to investigate the effects of adding very low doses of naltrexone to a methadone tapering treatment in opioid dependent individuals.

DETAILED DESCRIPTION:
Although many different techniques for opiate detoxification exist, the search continues for more effective approaches to reduce the duration and discomfort associated with opioid withdrawal. It has been shown that very low doses of naltrexone administered in the presence of opiates has analgesic and dependency reducing properties. The purpose of this study is to investigate the effects of very low doses of naltrexone administered during a methadone tapering schedule for opiate detoxification. In addition, this study will compare the effectiveness of two different dose regimens of naltrexone.

Participants in this double-blind study will be recruited among opioid dependent individuals already enrolled in a 6-day inpatient opioid detoxification program. Participants will be already receiving standard treatment to control discomfort during a methadone tapering schedule. Participants will be randomly assigned to one of three groups. Two of the groups will be given naltrexone; Group 1 will receive 0.125 mg each day, and Group 2 will receive 0.250 mg each day. Group 3 will receive a placebo. Participants will be evaluated upon enrollment for opiate addiction severity. They will continue to be evaluated daily for signs of withdrawal and salivary cortisol. An additional evaluation and urine test will be completed 1 day following discharge. Daily evaluations will take 15 minutes to complete. Seven days following discharge, participants will be contacted for a 20-minute phone interview. During the phone interview, participants will schedule an appointment to provide a final urine specimen for the detection of drugs of abuse.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV diagnosis of opiate dependence
* Reads and understands English

Exclusion Criteria:

* Serious medical disorders (e.g., uncontrolled hypertension, acute or chronic active hepatitis, kidney failure, uncontrolled diabetes)
* Psychiatric conditions that require intensive services (e.g., depression with suicidal ideation, psychosis)
* Mental retardation or other disorder that might limit ability to give informed consent
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2005-04; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Withdrawal intensity | 6 days

SECONDARY OUTCOMES:
Retention in treatment | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Mannelli, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Mannelli P, Wu LT, Peindl KS, Gorelick DA. Smoking and opioid detoxification: behavioral changes and response to treatment. Nicotine Tob Res. 2013 Oct;15(10):1705-13. doi: 10.1093/ntr/ntt046. Epub 2013 Apr 9. PMID 23572466
- [Derived] Mannelli P, Peindl K, Wu LT, Patkar AA, Gorelick DA. The combination very low-dose naltrexone-clonidine in the management of opioid withdrawal. Am J Drug Alcohol Abuse. 2012 May;38(3):200-5. doi: 10.3109/00952990.2011.644003. Epub 2012 Jan 10. PMID 22233189
- [Derived] Mannelli P, Peindl K, Patkar AA, Wu LT, Tharwani HM, Gorelick DA. Problem drinking and low-dose naltrexone-assisted opioid detoxification. J Stud Alcohol Drugs. 2011 May;72(3):507-13. doi: 10.15288/jsad.2011.72.507. PMID 21513688
- [Derived] Mannelli P, Peindl K, Patkar AA, Wu LT, Pae CU, Gorelick DA. Reduced cannabis use after low-dose naltrexone addition to opioid detoxification. J Clin Psychopharmacol. 2010 Aug;30(4):476-8. doi: 10.1097/JCP.0b013e3181e5c168. No abstract available. PMID 20631574
- [Derived] Mannelli P, Patkar AA, Peindl K, Gottheil E, Wu LT, Gorelick DA. Early outcomes following low dose naltrexone enhancement of opioid detoxification. Am J Addict. 2009 Mar-Apr;18(2):109-16. doi: 10.1080/10550490902772785. PMID 19283561